CLINICAL TRIAL: NCT03374722
Title: Opioid Withdrawal Symptoms in Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Suthinee Taesotikul, Principal investigator, Mahidol University
Other Study IDs: 10-60-68
Record Dates: First submitted 2017-12-12; First posted 2017-12-15 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Substance Withdrawal Syndrome; Critical Illness
MeSH Terms: conditions — Substance Withdrawal Syndrome; Critical Illness | interventions — Analgesics, Opioid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mechanically ventilated critically ill patients: Mechanically ventilated critically ill patients who receive opioid as continuous infusion for more than 24 hours
  Interventions: Drug: Opioids

INTERVENTIONS:
Drug: Opioids — Mechanically ventilated critically ill patients who receive continuous opioid infusion for more than 24 hours will be observed for withdrawal symptoms when rate of opioid infusion is disrupted or decreased

SUMMARY:
Most critically ill patients encounter pain and distress from acute illness, medical procedures and devices as well as routine care in the intensive care units (ICU). Opioids are principal analgesics that alleviate moderate to severe pain and facilitate patients to co-operate the course of treatment. However, prolong administration of opioids especially in mechanically ventilated patients can cause withdrawal symptoms if analgesics are rapidly weaning or acutely disruption. The opioid withdrawal symptoms (OWS) are well reported in critically ill children that cause discomfort and prolong weaning from mechanical ventilation. Weaning opioids and treatment of withdrawal symptoms are needed in order to decrease ventilator days, ICU and hospital length of stay. Conversely, there is lack of knowledge about incidence, clinical presentation, time course and appropriated assessment tool for withdrawal detection. Therefore, we conduct the study to explore an incidence of OWS, to identify factors associated OWS, to establish the assessment tool for OWS, and to report efficacy of the pharmacological treatment for OWS, in adult critically ill patients.

DETAILED DESCRIPTION:
The primary objective of the study is to explore incidence of OWS in adult critically ill patients. The secondary objectives are 1) to identify factor associated OWS, 2) establish the assessment tool for OWS for adults and 3) to report efficacy of the pharmacological treatment in OWS in adults patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* On mechanical ventilator at least 24 hours
* Received continuous infusion of opioid at least 24 hours
* Patient or legal surrogate who is willing and able to provide written informed consent and comply with all protocol requirements

Exclusion Criteria:

* Severely disturbed behavior pattern on account of underlying neurological disease (status epilepticus, encephalopathy, head trauma, brain injury, spinal cord injury)
* Preexisting psychiatric diagnosis
* Substance abuse prior to ICU admission
* Chronic alcohol drinking
* Pregnancy
* End-of-life care
* Death during ICU admission or during opioid IV infusion

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Intensive care units
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-10-07 (Actual)

PRIMARY OUTCOMES:
Incidence of opioid withdrawal symptoms | 0, 1, 3, 6, 24 and 72 hour after reduction or discontinuation of intravenous opioid
  Incidence of opioid withdrawal symptoms detected by self-developed assessment tool or the Diagnostic and Statistical Manual 5th edition (DSM-V)

SECONDARY OUTCOMES:
Weaning days | 28 days
  Time from initial weaning from mechanical ventilator until extubation
Ventilator days | 28 days
  Time from intubation until extubation
ICU length of stay | 28 days
  Time from admission to ICU until discharge from ICU

CONTACTS AND LOCATIONS:
Overall Officials: Suthinee Taesotikul, Pharm.D., Principal Investigator — Faculty of Pharmacy, Mahidol university
Locations (1):
- Faculty of Pharmacy, Mahidol University, Ratchathewi, Bangkok, Thailand

REFERENCES:
- [Result] Wang PP, Huang E, Feng X, Bray CA, Perreault MM, Rico P, Bellemare P, Murgoi P, Gelinas C, Lecavalier A, Jayaraman D, Frenette AJ, Williamson D. Opioid-associated iatrogenic withdrawal in critically ill adult patients: a multicenter prospective observational study. Ann Intensive Care. 2017 Sep 2;7(1):88. doi: 10.1186/s13613-017-0310-5. PMID 28866754
- [Result] Korak-Leiter M, Likar R, Oher M, Trampitsch E, Ziervogel G, Levy JV, Freye EC. Withdrawal following sufentanil/propofol and sufentanil/midazolam. Sedation in surgical ICU patients: correlation with central nervous parameters and endogenous opioids. Intensive Care Med. 2005 Mar;31(3):380-7. doi: 10.1007/s00134-005-2579-3. Epub 2005 Feb 16. PMID 15714323
- [Result] Brown C, Albrecht R, Pettit H, McFadden T, Schermer C. Opioid and benzodiazepine withdrawal syndrome in adult burn patients. Am Surg. 2000 Apr;66(4):367-70; discussion 370-1. PMID 10776874
- [Result] Cammarano WB, Pittet JF, Weitz S, Schlobohm RM, Marks JD. Acute withdrawal syndrome related to the administration of analgesic and sedative medications in adult intensive care unit patients. Crit Care Med. 1998 Apr;26(4):676-84. doi: 10.1097/00003246-199804000-00015. PMID 9559604
- [Derived] Taesotikul S, Dilokpattanamongkol P, Tangsujaritvijit V, Suthisisang C. Incidence and clinical manifestation of iatrogenic opioid withdrawal syndrome in mechanically ventilated patients. Curr Med Res Opin. 2021 Jul;37(7):1213-1219. doi: 10.1080/03007995.2021.1928616. Epub 2021 May 25. PMID 33966568